CLINICAL TRIAL: NCT04616300
Title: Cardiorespiratory Fitness, Inflammatory Biomarkers, and Cognitive Function Patterns During Treatment for Breast Cancer: a Prospective Cohort Study
Brief Title: Exercise and Cognitive (Brain) Function in Breast Cancer Patients Getting Chemotherapy After Breast Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Linda Trinh, Assistant Professor, University of Toronto
Other Study IDs: 38406
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: cardiorespiratory fitness; cognitive function; physical activity; chemotherapy treatment; cancer biomarkers
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will primarily identify longitudinal associations between cardiorespiratory fitness (CRF) and cognitive function pre- (baseline) to post-chemotherapy (~3 months). This will be a prospective study of 50 BCS. We hypothesize that breast cancer patients undergoing chemotherapy who have higher levels of CRF at baseline will have significantly improved measures of attention, executive function, and memory post-chemotherapy. In addition, the exploratory aims will examine the longitudinal associations between physical activity (PA) and cognitive function from pre- to post-chemotherapy and explore the associations between inflammatory and non-inflammatory biomarkers and CRF with cognitive function.

DETAILED DESCRIPTION:
Detailed Description:

Cognitive impairments are reported as a chief quality of life (QoL) complaint by approximately 75% of breast cancer survivors (BCS). Women who have undergone adjuvant chemotherapy are at the highest risk for cognitive impairments, that may affect BCS up to 20 years post-treatment.Despite the prevalence and significance, it is largely underdiagnosed and there are no proven treatments beyond symptom management. Several studies have assessed cognitive function in cancer populations. Increasing evidence highlights the role of lifestyle behaviours on cancer-related outcomes, ranging from QoL to prognosis. However, very few studies have examined the associations of lifestyle factors and cognitive function in BCS.One of the most important mediators of CRCI in BCS may be cardiorespiratory fitness (CRF).

Our overall objective is to examine the behavioral and biological mechanisms that contribute to cognitive decline in BCS undergoing chemotherapy using an epidemiologic, prospective cohort design.

Assessments taken at baseline (pre-chemotherapy) and post-chemotherapy (month 3). Cognitive Function will be assessed using the NIH toolbox cognition battery. Physical Activity. PA will be assessed by accelerometers and through self-report using the Godin-Leisure Time Exercise Questionnaire. Cardiorespiratory Fitness will be assessed using the 6-minute walk test to estimate maximum oxygen uptake (VO2max).Cancer Biomarkers will be assessed using venous blood (2 microtubes) will be drawn from the antecubital vein by a trained phlebotomist. Biological markers analyzed in blood will include a multiplex panel of inflammatory cytokines (i.e., IL1, IL6, TNFα), and brain-derived neurotrophic factor (BDNF).

Our proposed study will be instrumental in designing future targeted translational lifestyle interventions to improve cognitive health in BCS. In addition, understanding the trajectory of cognitive function as it relates to these factors will determine the opportune timeframe to intervene during the cancer care continuum for the greatest impact.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* histologically-confirmed stage I-III breast cancer, but prior to the initiation of chemotherapy (<1 cycle of adjuvant therapy or neoadjuvant therapy)
* no diagnosed major cognitive disorders and uncontrolled comorbidities.

Exclusion Criteria:

* received neoadjuvant chemotherapy and scheduled to receive adjuvant chemotherapy
* scheduled to receive concurrent radiation therapy with chemotherapy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 BCS from the Odette Cancer Centre and breast cancer organizations within the Greater Toronto Area
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Fluid Cognition (Composite) | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). This composite includes all the tests noted above that are fluid ability measures: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the normalized scores of each of the measures, and then deriving scale scores based on this new distribution. An Age-Adjusted Scale Score, Fully Adjusted Scale Score, Unadjusted Scale Score and Age-Adjusted National Percentile are provided for the Fluid Cognition Composite. The Fluid Cognition Composite is a more global assessment of individual and group fluid cognition functioning. Higher scores indicate higher levels of functioning.

SECONDARY OUTCOMES:
Executive/Attention | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Flanker Inhibitory Control and Attention Test tests the ability to inhibit visual attention to irrelevant task dimensions. A scoring algorithm integrates accuracy and reaction time yielding scores from 0 to 10. There are 40 trials and the average time to complete the task is 4 minutes.To interpret individual performance, one can evaluate all three types of scale scores in which higher scores indicate higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli.
Executive/Shifting | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Dimensional Change Card Sort Test involves a target visual stimulus that must be matched to 1 of 2 choice stimuli according to shape or color. Scoring is based on an algorithm that weights reaction time. A total of 40 trials require 4 minutes. Higher scores indicate higher levels of cognitive flexibility.
Working Memory | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The List Sorting Working Memory Test includes a series of stimuli is presented on the computer screen visually (object) and orally (spoken name), 1 at a time. Participants are instructed to repeat the stimuli to the tester in order of size, from smallest to largest. The List Sorting task takes approximately 7 minutes to administer. Test scores consist of total items correct across all trials. Higher scores indicate better working memory.The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Picture Vocabulary Test involves single words that are presented via an audio file, paired simultaneously with 4 screen images of objects, actions, and/or depictions of concepts. The participant will pick the picture that match
Episodic Memory | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Picture Sequence Memory Test involves a presentation of stimuli which are pictured objects and activities, thematically related but with no inherent order. For each trial, pictures appear in the center of the screen and then are moved 1 at a time into a fixed spatial order, as an audio file simultaneously describes the content of each. The score is based on the cumulative number of adjacent pairs of pictures remembered correctly over 3 learning trials. The test takes approximately 10 minutes. Higher scores indicate better episodic memory.
Language (oral reading) | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Oral Reading Recognition Test measures the ability to pronounce single printed words and/or to recognize letters. Items are administered by computer adaptive testing (CAT) and participant responses are entered by the tester. The CAT item bank contains approximately 250 items with only 30 to 40 that will be presented, depending on performance. Average administration time is 4 minutes. A higher Computed Score for Reading would mean that the participant is able to correctly identify more difficult words on the subsequent assessment, which may indicate developmental growth or a return to a previous level of functioning.
Language (picture vocabulary) | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Picture Vocabulary Test involves single words that are presented via an audio file, paired simultaneously with 4 screen images of objects, actions, and/or depictions of concepts. The participant will pick the picture that matches the spoken word. Total administration time is approximately 5 minutes. To interpret individual performance, one can evaluate all three types of scale scores. A participant's age-adjusted scale score at or near 100 indicates vocabulary ability that is average for the age level. Scores around 115 suggest above-average vocabulary ability, while scores around 130 suggest superior ability - in the top 2 percent nationally for age, based on Toolbox normative data.
Processing Speed (Pattern comparison) | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Pattern Comparison Processing Speed Test requires participants to identify whether two visual patterns are the "same" or "not the same." Average time of administration is 3 minutes and the score is the number of correct items (of a possible 130) completed in 90 seconds. Higher scores indicate faster speed of processing.
Crystallized Cognition | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). This composite includes the Picture Vocabulary and Reading Tests. This composite score is derived by averaging the normalized scores of each of the measures, and then deriving scale scores based on this 14 new distribution. An Age-Adjusted Scale Score, Fully Adjusted Scale Score, Unadjusted Scale Score and Age-Adjusted National Percentile are provided for the Crystallized Cognition Composite. Crystallized Cognition Composite is a more global assessment of individual and group verbal reasoning. Higher scores indicate higher levels of functioning.
Immediate Recall | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Auditory Verbal Learning Test (Rey) measures immediate recall. Unrelated words presented via audio recording and participant recalls as many as possible. he Rey is scored by taking the sum of the number of words recalled across all trials (possible range is 0-45 words). The raw score is most commonly used for interpretation of the Rey test, with higher scores reflecting better episodic memory.
Processing Speed (oral symbol digit test) | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Oral Symbol Digit Test measures speed of processing. Symbols on the screen are associated with a number, then presented with symbols without numbers. The Oral Symbol Digit Test is scored as the number of items answered correctly in 120 seconds (possible range is 0-144).Higher scores indicate better processing speed.
Objectively-assessed physical activity | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Objectively assessed PA was measured using Actigraph GTX3+ accelerometers (Pensacola, FL). Participants will wear the accelerometer on their non-dominant hip during waking hours for 7 consecutive days. Data will be downloaded in 60-s epochs and processed and converted to mean counts per minute in ActiLife software package (Version 6; Actigraph) to estimate daily minutes of light (101-1951 counts min-1), moderate (1952-5724 counts min-1), vigorous (≥ 5725 counts min-1), and total moderate-to-vigorous physical activity (MVPA; ≥ 1952 counts min-1) based on established cut-points (Freedson, Melanson, & Sirard, 1998). Estimated average daily minutes spent in each activity intensity category was calculated by dividing the number of minutes spent in each category by the total number of valid days worn.
Self-reported physical activity | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Physical activity will be assessed using a modified version of the validated leisure score index (LSI) from the Godin Leisure-Time Exercise Questionnaire (GLTEQ). Participants are asked to recall the average number of times per week and average duration they performed light (minimal effort, no perspiration), moderate (not exhausting, light perspiration), and vigorous (heart beats rapidly, sweating) physical activity during free time in the past month. The percentage of participants meeting the public health aerobic physical activity guidelines was calculated based on the physical activity guidelines recommended for cancer survivors by the American College of Sports Medicine. These guidelines recommend that individuals obtain 75 min of vigorous aerobic physical activity per week, 150 min of moderate aerobic physical activity per week, or an equivalent combination. Thus, will calculated physical activity minutes as moderate minutes plus two times the vigorous minutes.
Cancer biomarkers | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cancer Biomarkers will be assessed using venous blood (2 microtubes) will be drawn from the antecubital vein by a trained phlebotomist. Biological markers analyzed in blood will include a multiplex panel of inflammatory cytokines (i.e., IL1, IL6, TNFα), and brain-derived neurotrophic factor (BDNF).
Cardiorespiratory fitness | Change in from baseline (pre-chemotherapy) and post-chemotherapy (month 3).
  Cardiorespiratory Fitness will be assessed using the six-minute walk test (6MWT) to estimate maximum oxygen uptake (VO2max).The 6MWT measures the distance in meters an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes at their own pace.A lower score (reflecting less distance covered) indicates worse function.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre-Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellon SA, Ganz PA, Bower JE, Petersen L, Abraham L, Greendale GA. Neurocognitive performance in breast cancer survivors exposed to adjuvant chemotherapy and tamoxifen. J Clin Exp Neuropsychol. 2004 Oct;26(7):955-69. doi: 10.1080/13803390490510905. PMID 15742545
- [Background] Kesler SR, Kent JS, O'Hara R. Prefrontal cortex and executive function impairments in primary breast cancer. Arch Neurol. 2011 Nov;68(11):1447-53. doi: 10.1001/archneurol.2011.245. PMID 22084128
- [Background] Koppelmans V, Breteler MM, Boogerd W, Seynaeve C, Gundy C, Schagen SB. Neuropsychological performance in survivors of breast cancer more than 20 years after adjuvant chemotherapy. J Clin Oncol. 2012 Apr 1;30(10):1080-6. doi: 10.1200/JCO.2011.37.0189. Epub 2012 Feb 27. PMID 22370315
- [Background] Kesler S, Hadi Hosseini SM, Heckler C, Janelsins M, Palesh O, Mustian K, Morrow G. Cognitive training for improving executive function in chemotherapy-treated breast cancer survivors. Clin Breast Cancer. 2013 Aug;13(4):299-306. doi: 10.1016/j.clbc.2013.02.004. Epub 2013 May 4. PMID 23647804
- [Background] Von Ah D, Tallman EF. Perceived cognitive function in breast cancer survivors: evaluating relationships with objective cognitive performance and other symptoms using the functional assessment of cancer therapy-cognitive function instrument. J Pain Symptom Manage. 2015 Apr;49(4):697-706. doi: 10.1016/j.jpainsymman.2014.08.012. Epub 2014 Sep 18. PMID 25240787
- [Background] Frank JS, Vance DE, Triebel KL, Meneses KM. Cognitive Deficits in Breast Cancer Survivors After Chemotherapy and Hormonal Therapy. J Neurosci Nurs. 2015 Dec;47(6):302-12. doi: 10.1097/JNN.0000000000000171. PMID 26447567
- [Background] Von Ah D, Habermann B, Carpenter JS, Schneider BL. Impact of perceived cognitive impairment in breast cancer survivors. Eur J Oncol Nurs. 2013 Apr;17(2):236-41. doi: 10.1016/j.ejon.2012.06.002. Epub 2012 Aug 14. PMID 22901546
- [Background] Argyriou AA, Assimakopoulos K, Iconomou G, Giannakopoulou F, Kalofonos HP. Either called "chemobrain" or "chemofog," the long-term chemotherapy-induced cognitive decline in cancer survivors is real. J Pain Symptom Manage. 2011 Jan;41(1):126-39. doi: 10.1016/j.jpainsymman.2010.04.021. Epub 2010 Sep 15. PMID 20832978
- [Background] Jean-Pierre P, Johnson-Greene D, Burish TG. Neuropsychological care and rehabilitation of cancer patients with chemobrain: strategies for evaluation and intervention development. Support Care Cancer. 2014 Aug;22(8):2251-60. doi: 10.1007/s00520-014-2162-y. Epub 2014 Mar 27. PMID 24671433
- [Background] Zimmer P, Baumann FT, Oberste M, Wright P, Garthe A, Schenk A, Elter T, Galvao DA, Bloch W, Hubner ST, Wolf F. Effects of Exercise Interventions and Physical Activity Behavior on Cancer Related Cognitive Impairments: A Systematic Review. Biomed Res Int. 2016;2016:1820954. doi: 10.1155/2016/1820954. Epub 2016 Apr 10. PMID 27144158
- [Background] Wefel JS, Schagen SB. Chemotherapy-related cognitive dysfunction. Curr Neurol Neurosci Rep. 2012 Jun;12(3):267-75. doi: 10.1007/s11910-012-0264-9. PMID 22453825
- [Background] Ballard-Barbash R, Friedenreich CM, Courneya KS, Siddiqi SM, McTiernan A, Alfano CM. Physical activity, biomarkers, and disease outcomes in cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Jun 6;104(11):815-40. doi: 10.1093/jnci/djs207. Epub 2012 May 8. PMID 22570317
- [Background] Pierce JP, Stefanick ML, Flatt SW, Natarajan L, Sternfeld B, Madlensky L, Al-Delaimy WK, Thomson CA, Kealey S, Hajek R, Parker BA, Newman VA, Caan B, Rock CL. Greater survival after breast cancer in physically active women with high vegetable-fruit intake regardless of obesity. J Clin Oncol. 2007 Jun 10;25(17):2345-51. doi: 10.1200/JCO.2006.08.6819. PMID 17557947
- [Background] Zuniga KE, Mackenzie MJ, Roberts SA, Raine LB, Hillman CH, Kramer AF, McAuley E. Relationship between fruit and vegetable intake and interference control in breast cancer survivors. Eur J Nutr. 2016 Jun;55(4):1555-62. doi: 10.1007/s00394-015-0973-3. Epub 2015 Jun 30. PMID 26123915
- [Background] Jones LW, Haykowsky MJ, Swartz JJ, Douglas PS, Mackey JR. Early breast cancer therapy and cardiovascular injury. J Am Coll Cardiol. 2007 Oct 9;50(15):1435-41. doi: 10.1016/j.jacc.2007.06.037. Epub 2007 Sep 24. PMID 17919562
- [Background] Paterson DH, Cunningham DA, Koval JJ, St Croix CM. Aerobic fitness in a population of independently living men and women aged 55-86 years. Med Sci Sports Exerc. 1999 Dec;31(12):1813-20. doi: 10.1097/00005768-199912000-00018. PMID 10613433
- [Background] Klein RM. Inhibition of return. Trends Cogn Sci. 2000 Apr;4(4):138-147. doi: 10.1016/s1364-6613(00)01452-2. PMID 10740278
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Hartman SJ, Nelson SH, Myers E, Natarajan L, Sears DD, Palmer BW, Weiner LS, Parker BA, Patterson RE. Randomized controlled trial of increasing physical activity on objectively measured and self-reported cognitive functioning among breast cancer survivors: The memory & motion study. Cancer. 2018 Jan 1;124(1):192-202. doi: 10.1002/cncr.30987. Epub 2017 Sep 19. PMID 28926676
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Weller IM, Thomas SG, Gledhill N, Paterson D, Quinney A. A study to validate the modified Canadian Aerobic Fitness Test. Can J Appl Physiol. 1995 Jun;20(2):211-21. doi: 10.1139/h95-015. PMID 7640647
- [Background] Jones LW, Courneya KS, Mackey JR, Muss HB, Pituskin EN, Scott JM, Hornsby WE, Coan AD, Herndon JE 2nd, Douglas PS, Haykowsky M. Cardiopulmonary function and age-related decline across the breast cancer survivorship continuum. J Clin Oncol. 2012 Jul 10;30(20):2530-7. doi: 10.1200/JCO.2011.39.9014. Epub 2012 May 21. PMID 22614980
- [Background] Horowitz TS, Suls J, Trevino M. A Call for a Neuroscience Approach to Cancer-Related Cognitive Impairment. Trends Neurosci. 2018 Aug;41(8):493-496. doi: 10.1016/j.tins.2018.05.001. Epub 2018 Jun 12. PMID 29907436